CLINICAL TRIAL: NCT01939431
Title: Investigation of the Pathogenesis of Podoconiosis Using RNA-seq and Immunopathologic Approaches
Brief Title: Genetic and Other Aspects of Podoconiosis
Status: Terminated | Type: Observational
Why Stopped: Slow/Insufficient accrual
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913129; 13-HG-N129
Record Dates: First submitted 2013-09-05; First posted 2013-09-11 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Podoconiosis
Keywords: Podoconiosis; Ethiopian
MeSH Terms: conditions — Elephantiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (3):
- Advanced: advanced stage podoconiosis
- Control: non-podoconiosis controls
- Early: early stage podoconiosis

SUMMARY:
Background:

- Podoconiosis is a disease of the lymph vessels in the legs and feet. It is caused by long-term barefoot exposure to irritant soils, such as those in volcanic areas. It causes severe swelling and disfigurement, as well as infection and chronic pain. It mostly affects people who live in tropical Africa, Central and South America, and India. The reasons why some people develop this disease and others do not is not well understood. Researchers want to study people with the disease and healthy volunteers in Ethiopia. They will collect skin and blood samples to study genetic and other aspects of the disease.

Objectives:

- To collect skin and blood samples to study genetic and other aspects of podoconiosis.

Eligibility:

* Individuals at least 18 years of age who have podoconiosis (early stage or advanced stage).
* Healthy volunteers at least 18 years of age.
* Participants will be recruited from a study clinic and hospital in Ethiopia.

Design:

* Participants will be screened with a physical exam and medical history.
* Blood samples will be collected. A skin biopsy will be performed to collect tissue for study. People who have podoconiosis will provide affected and unaffected tissue. Healthy volunteers will provide a single skin biopsy sample.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
This research protocol is designed to study gene expression differentials and immunologic profile and histopatologic presentation of podoconiosis by comparing cases and controls in Ethiopia. Podoconiosis is a geochemical lymphedema of the lower limbs resulting from long term barefoot exposure to irritant red clay soils of volcanic origin. The disease imposes huge social and economic burden and affects more than 4 million individuals in tropical Africa, Central and South America, and North India. The pathologic changes in podoconiosis are still not known and the histopathologic features of the disease have not been well studied. Our recent genome-wide association study revealed that variants in HLA class II genes (HLA-DRB1, -DQB1, and -DQA1) are associated with podoconiosis, and suggests that the disease may be a Tcell mediated inflammatory condition (New Eng J Med 2012). The objectives of the present study are to investigate the immunologic profiles and gene expression differences between podoconiosis patients and healthy controls. The study will include 150 subjects consisting of 100 cases (50 early stage and 50 advanced stage), and 50 controls from Ethiopia. Anonymized discarded skin tissue samples will be obtained from excised nodules of 50 advanced stage patients that undergo nodulectomy (surgical excisions of nodules) in Bahir Dar Hospital. Punch biopsies will be obtained from affected skin tissues (epidermis and dermis) of 50 early stage podoconiosis patients that attend routine treatment in Dur-Bete

Podoconiosis Center, and normal skin tissues (epidermis and dermis) of 50 control subjects undergoing orthopedic surgery of the lower legs in Bahir Dar Hospital. We will also obtain 6 mm skin tissue punch biopsies from the unaffected areas in the lower limbs of all podoconiosis patients and peripheral blood samples (PBS) from all study subjects. RNA from PBS and T cells separated from other cells will be extracted in Armauer Hansen Research Institute of Ethiopia (AHRI) and will be shipped along with skin biopsies that will be kept in liquid nitrogen to CRGGH/NHGRI. Back-up samples will be kept in AHRI. We will use RNA-seq, a high throughput RNA sequencing technology, to characterize the transcriptome by sequencing complementary DNAs (cDNAs) followed by mapping of the sequence reads to the genome. Generation of double-stranded cDNA from mRNA and quantitation of cDNA concentration will

be done in our lab at NIH. Sequencing will be done by a commercial high throughput sequencing company, SeqWright (Houston, TX) an Illumina certified service provider. Immunologic profiling will be done using a FACSCalibur type flow cytometry. Analysis of data will be done using appropriate statistical programs and pipeline suites as described below. This study is expected to reveal differential gene expression between podoconiosis patients and controls. Furthermore, it will chart the evolution of gene expression signatures in podoconiosis patients through the different clinical stages of the disease. The findings could potentially lead to biomarkers that complement the clinical and genetic characteristics of the disease. The histopathological studies will provide a rich description of cutaneous and immunologic response across the spectrum of the disease. The integration of clinical, immunological, genetic, cellular and molecular characteristics of the disease will facilitate the development of a model for the natural history and pathogenesis of this neglected tropical disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All individuals included in our study will be adults (greater than or equal to 18 years) because the average age of onset of the disease is during the third decade of life. In addition, in Ethiopia the legal age to give independent consent for research is 18 years or older. Previous studies have shown that diagnosis of podoconiosis using physical diagnostic criteria in endemic highland areas is highly accurate. To rule out filarial elephantiasis, a rapid ICT card test will be done. Advanced stage podoconiosis cases will be included in the study based on prior assessment of an experienced surgeon (Dr Wendemagegn Enbiale Yeshanehe) who assures eligibility for nodulectomy if a patient with clinical stage III, IV or V podoconiosis has fibrotic nodules. Early clinical stage podoconiosis patients will be individuals with negative filarial test and at clinical stages I or II. Controls will be individuals with no past or current history, signs and symptoms of podoconiosis and no family history of podoconiosis.

EXCLUSION CRITERIA:

-In addition to clinical criteria that make patients and controls non-eligible to undergo surgery, we will also exclude individuals with skin infection, skin lesion at the prospective biopsy site, medical contradictions to biopsy, history of adenolymphangitis during the previous 2 weeks, topical steroid treatment during the previous 2 weeks, with biologically related family members that are included in the study, recent infection, use of systemic antibiotics and use of systemic steroids. Attempts will be made to enroll an equal number of men and women. No prisoners, pregnant women or fetuses will be included in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with podoconiosis@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Natural History | Ongoing
  To study genetic and other aspects of podoconiosis using data from skin and blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Rotimi, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- Bahir Dar University, Medical and Healath Science College, Bahir Dar, Ethiopia

REFERENCES:
- [Background] Bullard JH, Purdom E, Hansen KD, Dudoit S. Evaluation of statistical methods for normalization and differential expression in mRNA-Seq experiments. BMC Bioinformatics. 2010 Feb 18;11:94. doi: 10.1186/1471-2105-11-94. PMID 20167110
- [Background] Cheng WC, Shu WY, Li CY, Tsai ML, Chang CW, Chen CR, Cheng HT, Wang TH, Hsu IC. Intra- and inter-individual variance of gene expression in clinical studies. PLoS One. 2012;7(6):e38650. doi: 10.1371/journal.pone.0038650. Epub 2012 Jun 18. PMID 22723873
- [Background] Davey G, Gebrehanna E, Adeyemo A, Rotimi C, Newport M, Desta K. Podoconiosis: a tropical model for gene-environment interactions? Trans R Soc Trop Med Hyg. 2007 Jan;101(1):91-6. doi: 10.1016/j.trstmh.2006.05.002. Epub 2006 Aug 1. PMID 16884751